CLINICAL TRIAL: NCT06575842
Title: Accuracy of Continuous Glucose Monitors During the Perioperative Period in Youth With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 24-0717
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
Keywords: Anesthesia; Continuous glucose monitors; Accuracy; Pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing anesthesia: Pediatric patients who are undergoing a surgical procedure with anesthesia. Patients will have type 1 diabetes and be wearing a continuous glucose monitor as part of routine care.

SUMMARY:
This study is assessing the accuracy of continuous glucose monitors during surgical procedures requiring anesthesia.

DETAILED DESCRIPTION:
This study is an observational study design that includes collection of continuous glucose data and venous blood glucose data (from either an IV or fingerstick) from a blood glucose meter. All subjects will be undergoing a surgical procedure that requires anesthesia. The primary outcome of this study is to evaluate the accuracy of the CGM glucose values in comparison to the reference glucometer glucose value during anesthesia. There is currently limited data on accuracy of CGMs during these events and therefore it is not know whether CGM glucose data is reliable to be used as the sole source of glucose monitoring during surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 2 to 26 years of age at the time of enrollment.
2. Participants will have a diagnosis of type 1 diabetes on insulin therapy and requiring close glucose monitoring during the hospitalization and the perioperative period.
3. Participant currently wearing a continuous glucose monitor (for example: Dexcom G6 or G7; Freestyle Libre 2, 2 Plus, or 3; Medtronic Guardian 3 or 4; or future sensors as they become available) for home diabetes management and willing to share personal CGM data with the BDC clinical CGM account.

Exclusion Criteria:

1. Pregnancy.
2. Currently using hydroxyurea.
3. A condition that the investigator determines would prevent the patient from participation.

Ages: 2 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants will have a clinical diagnosis of type 1 diabetes and be wearing a continuous glucose monitor as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CGM compared to blood glucose using standard statistical methods including mean absolute relative difference (MARD). | Perioperatively (length of time will vary based on the operative procedure)
  Accuracy assessment will be completed comparing CGM glucose values to blood glucose values using standard statistical assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided